CLINICAL TRIAL: NCT06999720
Title: A Phase I, Randomized, Double-Blinded, Placebo-Controlled, Single Dose and Multiple Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Pharmacodynamics of HX15001 in Adult Healthy Volunteers.
Brief Title: Study of HX15001 in Adult Healthy Volunteers.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Helixon Biotechnology (Suzhou) Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HXN-IMM-001-I
Record Dates: First submitted 2025-05-22; First posted 2025-05-31 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sagittal Abdominal Diameter; mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A - Single-Ascending Dose (SAD) (Experimental): Participants will receive a single intravenous dose of HX15001 (Cohort 1-7).
  Interventions: Drug: HX15001 (SAD)
- Placebo SAD Cohorts (1-7) (Placebo Comparator): Participants will receive multiple intravenous dose of Placebo
  Interventions: Drug: Placebo
- Part B - Multiple Ascending Dose (MAD) (Experimental): Participants will receive multiple intravenous doses of HX15001 (Cohort 8-9).
  Interventions: Drug: HX15001 (MAD)
- Placebo MAD Cohorts (8-9) (Placebo Comparator): Participants will receive multiple intravenous dose of Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HX15001 (SAD) — Part A (Single Ascending Dose), participants will receive a single intravenous dose of HX15001 at escalating dose levels in sequential cohorts (Cohorts 1-7).
  Arms: Part A - Single-Ascending Dose (SAD)
Drug: Placebo — Participants will receive matching placebo across cohorts 1-7 of the study.
  Arms: Placebo SAD Cohorts (1-7)
Drug: HX15001 (MAD) — In Part B (Multiple Ascending Dose), participants will receive multiple intravenous doses of HX15001 in cohorts 8 and 9 to assess safety, tolerability, and pharmacokinetics.
  Arms: Part B - Multiple Ascending Dose (MAD)
Drug: Placebo — Participants will receive matching placebo across cohorts 8-9 of the study.
  Arms: Placebo MAD Cohorts (8-9)

SUMMARY:
This is a phase I, randomized, double-blinded, placebo-controlled, single and multiple dose escalation study to evaluate the safety, tolerability, pharmacokinetic characteristics and pharmacodynamics of HX15001 in adult healthy participants.

The study consists of two parts: Part A involves single-dose escalation (Cohorts 1-7), and Part B involves multiple-dose escalation (Cohorts 8-9).

The primary objective of this study is to characterize the safety and tolerability of single and multiple doses of HX15001 in healthy subjects.

DETAILED DESCRIPTION:
This study consists of two parts. Part A: This part includes seven sequential ascending-dose cohorts, designated as Cohorts 1 through 7. Cohort 1 and Cohort 6 will enroll four healthy subjects in each cohort. Cohort 2 will enroll six healthy subjects. The remaining four cohorts will enroll eight healthy subjects each.

On Day 1, after final eligibility has been determined, subjects in Cohorts 1-5 will be randomly assigned to receive a single subcutaneous dose (which may be split into multiple dosing syringes) of HX15001 or placebo, while subjects in Cohorts 6 and 7 will be randomly assigned to receive a single intravenous infusion of HX15001 or placebo. The doses for Cohorts 1-7 will be administered as per the protocol.

Part B: This part consists of two multiple-dose cohorts (Cohorts 8 and 9), each enrolling eight healthy subjects. Subjects in these cohorts will receive subcutaneous doses of HX15001 or placebo on Days 1, 15, and 43. Dosing will be followed by safety, pharmacokinetic, pharmacodynamic, and immunogenicity assessments.

Study Period Part A: Screening：Up to 28 days Treatment：Day 1 single dose Follow up: 112 days including Day 1 (Cohort 1-3) 140 days including Day 1 (Cohort 4-7) Part B: Screening：Up to 28 days Treatment：Day 1, Day 15, Day 43 (single dose on each visit) Follow up: 20 weeks (Day 183) The final follow-up visit will be determined based on the safety and PK data derived from the previous SAD and MAD cohorts, which may be earlier or later than Day 183 (±7 days

ELIGIBILITY:
Inclusion Criteria:

1. An informed consent document signed and dated by the subject.
2. Healthy male and female subjects of any ethnic origin between the ages of 18 and 55 years, inclusive.
3. Have a Body mass index (BMI) of 18-32 kg/m2 , inclusive; with body weight ≥50 kg during the screening.
4. In good health, as determined by the investigator at Screening procedures, with no clinically significant findings from medical history, physical examination, 12-lead ECG, vital signs measurements, and clinical laboratory evaluations.
5. Subjects must be willing to understand and comply with all research procedures and restrictions, and able to communicate effectively with researchers.

Exclusion Criteria:

1. Females who are pregnant, planning to become pregnant, or breastfeeding during the trial.
2. Has a positive result of pregnancy test at Screening or Baseline
3. History of HIV infection, hepatitis B, hepatitis C or syphilis; positive testing for HIV, hepatitis B, HCV Ab or serological reaction of syphilis
4. Subjects at risk for tuberculosis (TB).
5. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol;
6. Has received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 30 days or 5 half-lives prior to dosing, or plan to receive another experimental agent during the duration of this trial;
7. Subjects who have donated blood (excluding plasma donations) of approximately 1 pint (500 mL) or more within 30 days prior to dosing, or those who plan to donate blood during the study period or within 30 days after the end of the study;
8. Use of prescription or over-the-counter drugs or dietary or herbal supplements within 7 days or 5 half-lives (whichever is longer) prior to dosing
9. Triplicate 12-lead electrocardiogram (ECG) that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
10. Has clinically significant interventional therapies (surgery, paracentesis, etc.) within 6 months prior to dosing, or plan to have any surgeries during the duration the trial.
11. History of any hypersensitivity or allergic reaction to drugs;
12. Has any other conditions that would, in the opinion of the investigator, put the subjects at increased risk for participation in this trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) cohort 1-3 | Up to day 113
  Incidence, severity, and causal relationship of Serious Adverse Events (SAEs) including changes in laboratory parameters (Hematology, Chemistry panels, Coagulation and Urinalysis); 12-lead ECGs parameters; Vital signs (Blood pressure, heart rate, respiratory rate and body temperature)
Adverse Events (AEs) and Serious Adverse Events (SAEs) cohort 4-7 | Up to day 141
  Incidence, severity, and causal relationship of Serious Adverse Events (SAEs) including changes in laboratory parameters (Hematology, Chemistry panels, Coagulation and Urinalysis); 12-lead ECGs parameters; Vital signs (Blood pressure, heart rate, respiratory rate and body temperature)
Adverse Events (AEs) and Serious Adverse Events (SAEs) cohort 8-9 | Up to day 183
  Incidence, severity, and causal relationship of Serious Adverse Events (SAEs) including changes in laboratory parameters (Hematology, Chemistry panels, Coagulation and Urinalysis); 12-lead ECGs parameters; Vital signs (Blood pressure, heart rate, respiratory rate and body temperature)

SECONDARY OUTCOMES:
Cmax | Up to day 113 (cohort 1-3) Up to day 141 (Cohort 4-7) Up to day 183 (Cohort 8-9)
  Maximum concentration after single and multiple ascending doses
Tmax | Up to day 113 (cohort 1-3) Up to day 141 (Cohort 4-7) Up to day 183 (Cohort 8-9)
  Time to reach maximum concentration after single and multiple ascending doses
t1/2 | Up to day 113 (cohort 1-3) Up to day 141 (Cohort 4-7) Up to day 183 (Cohort 8-9)
  Half life after single and multiple ascending doses
AUC | Up to day 113 (cohort 1-3) Up to day 141 (Cohort 4-7) Up to day 183 (Cohort 8-9)
  Area under the curve after single and multiple ascending doses
ADA | Up to day 113 (cohort 1-3) Up to day 141 (Cohort 4-7) Up to day 183 (Cohort 8-9)
  Incidence of anti-drug antibody after single and multiple ascending doses

CONTACTS AND LOCATIONS:
Locations (1):
- Q-Pharm Pty Ltd., Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No